CLINICAL TRIAL: NCT05992727
Title: Evaluation of Galectin 3 Level in Serum and Saliva of Pemphigus Patients and Its Correlation With Disease Severity and Systemic Comorbidities
Brief Title: Evaluation of Galectin-3 in Serum and Saliva of Pemphigus Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Fathy Ahmed, Doctor, Assiut University
Other Study IDs: Galectin -3 and pemphigus
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Galectin-3 and Pemphigus
MeSH Terms: conditions — Pemphigus | interventions — Blood Cell Count; Kidney Function Tests; Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1( cases): Galectin 3 will be measured in 30 Patients who are with active stage of pemphigus either newly diagnosed or in a relapse. The diagnosis of each patient is based on clinical examination and histopathological examination.
  Interventions: Diagnostic Test: Galectin 3 measurement in serum and saliva by ELIZA
- Group 2( controls): Galectin 3 will be measured in30 age and sex matched healthy controls
  Interventions: Diagnostic Test: Galectin 3 measurement in serum and saliva by ELIZA

INTERVENTIONS:
Diagnostic Test: Galectin 3 measurement in serum and saliva by ELIZA — Galectin 3 measurement in serum and saliva by ELISA in the two groups
  Other Names: complete blood count,renal function tests, random blood sugar,urine analysis and echocardiography

SUMMARY:
Assessment of the expression of galectin-3 in serum and saliva of pemphigus patients and compare it with age and sex matched controls. We want to detect whether a correlation exists between galectin-3 level in serum, as well as saliva and disease activity score by Autoimmune Bullous Skin Disorder Intensity Score (ABSIS).

DETAILED DESCRIPTION:
Pemphigus is a potentially life- threatening immune mediated bullous disease that affects the skin and mucous membranes with a significant impact on quality of life (1). It is due to production of autoantibodies against desmogleins (adhesion molecules of the epidermis) leading to disruption of junctions between keratinocytes and subsequently acantholysis (2).

Pemphigus diseases are classified based on the clinical, histopathological features, as well as on the specific antigens against which the autoantibodies are produced. The main forms are pemphigus vulgaris (PV) and pemphigus folia¬ceus (PF), but other non-classical forms of pemphigus have also been described as paraneoplastic pemphigus, pemphigus herpetiformis, and IgA pemphigus (3). PV is the main clinical form of pemphigus, accounting for approximately 70% of cases; it is also considered the most severe form of the disease (4).

IgG is the main immunoglobulin seen along the dermal-epidermal junction in pemphigus patients, in addition most patients generate IgE autoantibody response. Soluble CD23 and galectin-3 are the two main elements of the IgE (5).

Galectin-3(Gal-3) is a beta galactoside-binding lectins that is essential in the cell-to-cell or matrix adhesion, as well as plays an important role in cell growth, differentiation, macrophage activation, antimicrobial activity, angiogenesis, and apoptosis. It broadly exists in the nucleus and cytoplasm of various cell types or may be found extracellularly on the cell surface (6) .Gal-3 is readily secreted to the cell surface and into biological fluids as serum, urine, tears and saliva from injured and inflammatory cells. So, it can be used as a sensitive diagnostic or prognostic biomarker for various pathological conditions (7).

Gal-3 has been used as a novel biomarker in the early detection of myocardial dysfunction and heart failure. Many cardiac biomarkers which reflect cardiac inflammation and fibrosis may also contribute to the progression of kidney disease (8, 9) A previous study reported a significant decrease in galectin-3 cytoplasmic and nuclear expression around blisters compared with adjacent unaffected skin in PV, which may play a role in extension of acantholysis (5). To the best of our knowledge, no previous studies assessed the role of Gal-3 in serum or saliva of pemphigus patients.

ELIGIBILITY:
Inclusion Criteria:

Patients with active stage of pemphigus.

Exclusion Criteria:

1. Patients who were on topical ttt, systemic corticosteroids or other immunosuppressive drugs in the last one month.
2. Patients with disease attack duration more than 1 week.
3. Patients with any other concomitant dermatological or chronic systemic diseases.

   -

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pemphigus patients in active stage either newly diagnosed or in a relapse. The diagnosis of each patient is based on clinical examination , histopathological examination and direct immunofluorescence.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-08-08 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Galectin 3 | 1 year
  Three millimeters of blood will be withdrawn aseptically from all patients and controls from the antecubital vein using disposable plastic syringe. The sera will be separated and stored at -20 C. Saliva will be collected from patients and controls after asking them to refrain from eating and drinking (except for water) for 2 hours before collection. Then, they will be asked to rinse their mouth with water, tilt their heads down, pool saliva in the mouth for 1 minute, drool into a sterile falcon tube. Saliva will be separated and stored also at-20 C. Human Gal-3 ELISA kit will be used for quantitative measurement of serum and saliva Gal-3 levels. The assay will be performed according to the manufacturer's instructions.
Develop a novel biomarker in serum and saliva of pemphigus patients and to detect its correlation with disease activity, as well as systemic comorbidities. | 1year
  All patients will be subjected to complete history taking, meticulous general, dermatological examination and routine investigations. Echocardiography, kidney function tests and urine analysis will be conducted for all the participants. Disease severity will be assessed by ABSIS score with a maximum score of 206. It uses the rule of 9s to assess the percentage of involvement of blisters and erosions on the skin combined with a weighting factor for the stage of the blistering and erosions. Oral involvement is based on 2 scores comprising the extent (presence of lesions) and severity (discomfort during eating and drinking)

REFERENCES:
- [Result] Aghighi M, Pukhalskaya T, Smoller BR. Immunohistochemical Expression of Galectin-3 in Pemphigus Vulgaris. Am J Dermatopathol. 2021 Dec 1;43(12):e165-e168. doi: 10.1097/DAD.0000000000001939. PMID 33767069